CLINICAL TRIAL: NCT04347486
Title: Pharmacokinetic-pharmacodynamic Analysis of Conventional Reversal of Rocuronium-induced Neuromuscular Blockade by Sugammadex in Children
Brief Title: Pharmacokinetic-pharmacodynamic Analysis of Sugammadex for Conventional Reversal in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Principal Investigator, Hee-Soo Kim, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2002-148-1105
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Anesthesia, General; Neuromuscular Blockade
Keywords: Sugammadex; Pharmacokinetics; Pharmacodynamics; Pediatric anesthesia
MeSH Terms: interventions — Sugammadex; Atropine; Neostigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Sugammadex 2mg (Experimental): Administer 2mg/kg of sugammadex on reappearance of T2 by Train-of-Four stimulation
  Interventions: Drug: Sugammadex Injection 2mg/kg
- Sugammadex 4mg (Experimental): Administer 4mg/kg of sugammadex on reappearance of T2 by Train-of-Four stimulation
  Interventions: Drug: Sugammadex Injection 4mg/kg
- Sugammadex 8mg (Experimental): Administer 8mg/kg of sugammadex on reappearance of T2 by Train-of-Four stimulation
  Interventions: Drug: Sugammadex Injection 8mg/kg
- Conventional reversal (Active Comparator): Administer conventional neuromuscular reversal agent (0.02mg/kg of atropine and 0.03mg/kg of neostigmine) on reappearance of T2 by Train-of-Four stimulation
  Interventions: Drug: Neuromuscular reversal agent injection

INTERVENTIONS:
Drug: Sugammadex Injection 2mg/kg — Intravenous injection of 2mg/kg of sugammadex sodium on reappearance of T2
  Other Names: Bridion 2mg/kg
  Arms: Sugammadex 2mg
Drug: Sugammadex Injection 4mg/kg — Intravenous injection of 4mg/kg of sugammadex sodium on reappearance of T2
  Other Names: Bridion 4mg/kg
  Arms: Sugammadex 4mg
Drug: Sugammadex Injection 8mg/kg — Intravenous injection of 8mg/kg of sugammadex sodium on reappearance of T2
  Other Names: Bridion 8mg/kg
  Arms: Sugammadex 8mg
Drug: Neuromuscular reversal agent injection — Intravenous injection of 0.02mg/kg of atropine and 0.03mg/kg of neostigmine
  Other Names: Atropine and neostigmine
  Arms: Conventional reversal

SUMMARY:
This study administers sugammadex sodium to pediatric patients under general anesthesia with rocuronium. Pharmacokinetic and pharmacodynamic analysis are performed based on plasma concentration of sugammadex sodium and monitoring of neuromuscular blockade.

DETAILED DESCRIPTION:
This study enrolls pediatric patients undergoing surgery under general anesthesia with need for reversal of neuromuscular blockade, aged between 2 and 18 years old.

After routine anesthetic induction with 1% propofol and 0.6mg/kg of rocuronium, maintenance of anesthesia with total intravenous anesthesia is commenced. For neuromuscular monitoring, train-of-four (TOF) count and T4/T1 ratio are monitored, with recording of the time to recovery of the T4/T1 ratio to 0.7, 0.8 and 0.9.

On reappearance of T2 after rocuronium administration , 2 or 4 or 8mg/kg of sugammadex sodium or conventional neuromuscular reversal agent is administered according to randomization table.

For pharmacokinetic analysis, patient blood sample is obtained before / 2 min after rocuronium administration, before / 2min / 5min / 15min / 60min / 120min / 240min / 480min after sugammadex administration. Plasma concentration of rocuronium and sugammadex sodium are analyzed via high-performance liquid chromatography with mass spectrometric detection.

ELIGIBILITY:
Inclusion Criteria:

* All of below Pediatric patients undergoing surgery under general anesthesia with requirement of early reversal of neuromuscular blockade Aged between 2 and 17 American Society of Anesthesiologists Physical Status Classification 1 and 2

Exclusion Criteria:

* Any of below One or more legal guardian declines to enroll in the study History of hypersensitivity to any anesthetic agents including rocuronium Presence of underlying cardiovascular or genitourinary disease Under usage of neuromuscular blocking agents before surgery Under usage of drugs influencing the effect of neuromuscular blocking agents History of malignant hyperthermia Anticipation of massive hemorrhage during surgery

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Neuromuscular recovery | up to 30 minutes to 1 hour
  Time to recovery of train-of-four T4/T1 ratio to 90% after sugammadex sodium or neuromuscular reversal agent administration up to 30 minutes to 1 hour.

SECONDARY OUTCOMES:
Plasma concentrations | From anesthetic induction to 480 minutes after sugammadex administration
  Plasma concentrations of rocuronium and sugammadex sodium

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gijsenbergh F, Ramael S, Houwing N, van Iersel T. First human exposure of Org 25969, a novel agent to reverse the action of rocuronium bromide. Anesthesiology. 2005 Oct;103(4):695-703. doi: 10.1097/00000542-200510000-00007. PMID 16192761
- [Background] Sorgenfrei IF, Norrild K, Larsen PB, Stensballe J, Ostergaard D, Prins ME, Viby-Mogensen J. Reversal of rocuronium-induced neuromuscular block by the selective relaxant binding agent sugammadex: a dose-finding and safety study. Anesthesiology. 2006 Apr;104(4):667-74. doi: 10.1097/00000542-200604000-00009. PMID 16571960
- [Background] Sparr HJ, Vermeyen KM, Beaufort AM, Rietbergen H, Proost JH, Saldien V, Velik-Salchner C, Wierda JM. Early reversal of profound rocuronium-induced neuromuscular blockade by sugammadex in a randomized multicenter study: efficacy, safety, and pharmacokinetics. Anesthesiology. 2007 May;106(5):935-43. doi: 10.1097/01.anes.0000265152.78943.74. PMID 17457124
- [Background] Ploeger BA, Smeets J, Strougo A, Drenth HJ, Ruigt G, Houwing N, Danhof M. Pharmacokinetic-pharmacodynamic model for the reversal of neuromuscular blockade by sugammadex. Anesthesiology. 2009 Jan;110(1):95-105. doi: 10.1097/ALN.0b013e318190bc32. PMID 19104176
- [Background] Won YJ, Lim BG, Lee DK, Kim H, Kong MH, Lee IO. Sugammadex for reversal of rocuronium-induced neuromuscular blockade in pediatric patients: A systematic review and meta-analysis. Medicine (Baltimore). 2016 Aug;95(34):e4678. doi: 10.1097/MD.0000000000004678. PMID 27559972
- [Derived] Ji SH, Huh KY, Oh J, Jeong HJ, Jang YE, Kim EH, Lee JH, Kim JT, Kim HS. Conventional reversal of rocuronium-induced neuromuscular blockade by sugammadex in Korean children: pharmacokinetics, efficacy, and safety analyses. Front Pharmacol. 2023 Apr 13;14:1127932. doi: 10.3389/fphar.2023.1127932. eCollection 2023. PMID 37124204